CLINICAL TRIAL: NCT01106053
Title: An Exploration of the Effects of the Dopamine Agonist Pramipexole on Binge Antecedants, Binge Frequency, and Weight in Binge Eating Disorder
Brief Title: Pramipexole for Binge Eating Disorder
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants were recruited and study has been closed.
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Reseach Scientist, Neuropsychiatric Research Institute, Fargo, North Dakota
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEDA-Pramipexole
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Binge Eating Disorder
Keywords: Binge eating disorder; Food craving; Obesity; Pramipexole; Mirapex; Binge
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pramipexole (Experimental): Open-label trial of pramipexole.
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole — Pramipexole tablet titrated up to a maximum dosage of 0.5 mg three times daily (1.5 mg/day).
  Other Names: Mirapex

SUMMARY:
This study is being conducted to evaluate the effects that the drug pramipexole has on mood, food craving, and other behaviors that may be related to binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-50 years
* Women of child-bearing potential and males must agree to practice an accepted method of birth control. All women must have a negative pregnancy test at baseline.
* Good general health as demonstrated by history and physical examination.
* Body mass index of 30 kg/m2 or higher at the screening visit.
* Meet criteria for binge eating disorder as assessed through the SCID-1 and EDE.

Exclusion Criteria:

* Subjects with any unstable medical condition, or any current or past medical condition which in the opinion of the study physician and/or the principal investigator may increase the risks associated with pramipexole and study participation. Medical appropriateness will be determined through history and physical exam.
* Subjects with any current Axis I psychiatric diagnosis as determined through the Structured Clinical Interview for DSM-IV for Axis I disorders (SCID-1) interview (aside from BED).
* Subjects with a Hamilton Depression Rating Scale score greater than or equal to 12 at the screening visit.
* Subjects who report any history of hallucinations or delusions.
* Participants taking an antidepressant or other regularly used psychotropic medication which may confound the study results
* Subjects with any current or history of an impulse control spectrum disorder, other than binge eating disorder,(such as pathological gambling, compulsive shopping, etc.) at screening as determined by the Structured Clinical Interview for DSM-IV Impulse Control Module.
* Subjects with any history of suicide attempts or current suicidal ideations.
* Subjects that have used tobacco products on a routine basis within the past six months.
* Subjects enrolled in any formal treatment programs or research protocols for binge eating disorder at present, or within the past 30 days.
* Subjects routinely taking any medication known to produce weight change (ex. olanzapine, amitriptyline, steroid medications, etc., other than oral contraceptives, stable thyroid replacement drugs, etc.), or medications with drug-drug interactions with pramipexole.
* Subjects who are currently breast-feeding.
* Subjects who have participated in an investigational drug trial in the past 30 days.
* Subjects who meet DSM IV-TR criteria for alcohol or drug abuse in the past year.
* Subjects with an allergy to pramipexole or tablet constituents.
* Subjects with hepatic dysfunction as determined through a hepatic panel obtained at the screening visit.
* Subjects with an elevated blood pressure or pulse at screening (140/90 mmHg or above or pulse of greater than 100 beats/minute after being seated and stationary for at least five minutes, or as determined at the discretion of the study physician and/or principal investigator) or history of serious cardiac events (myocardial infarction, arrhythmia, stroke, etc).
* Subjects with a history of renal dysfunction or with a creatinine clearance of less than 60 ml/min based upon a serum creatinine obtained during screening and as calculated with the Cockroft and Gault equation.
* Subjects with a positive urine drug screen.
* Any participant with Parkinson's disease or symptoms suggestive of probable Parkinson's disease.
* Subjects who have an Epworth Sleep Scale (ESS) score of >7 at screening. ESS scores > 7 have been associated with an increased risk of sleep attacks (Plowman et al., 2005).
* Any participant who demonstrates clinically significant orthostatic blood pressure changes or is symptomatic during the screening visit, as defined under "orthostatic blood pressure monitoring."
* History of bariatric surgery.
* Participants who report a history of obstructive sleep apnea, excessive fatigue, or any sleep disorder which in the opinion of the principal investigator or study medical personnel would increase the participant's risk of experiencing excessive somnolence with pramipexole.
* Participant has had a change in medication regimen in the last month (dose, starting a new medication, or stopping a medication).
* Participant is employed by, or has an immediate family member employed by NRI.
* Participant has participated in a formal weight loss program in the last month (e.g. Weight Watchers, Jenny Craig, etc.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Frequency of binge eating | Baseline followed by weekly during the seven week protocol

SECONDARY OUTCOMES:
Body weight | Baseline followed by weekly during the seven week protocol
Frequency and extent of craving for food using validated instruments | Baseline followed by weekly during the seven week protocol
Assessment of mood ratings using a validated instrument | Baseline followed by weekly during the seven week protocol

CONTACTS AND LOCATIONS:
Overall Officials: Kristine J Steffen, PharmD, PhD, Principal Investigator — Neuropsychiatric Research Institute, Fargo, ND

REFERENCES:
- See also: NRI website — http://www.nrifargo.com